CLINICAL TRIAL: NCT00463060
Title: Phase I/II Study of Stereotactic Radiation Therapy and Concurrent and Adjuvant Sutent (SU11248) as Treatment for Oligometastatic Disease
Brief Title: Sutent and Radiation as Treatment for Limited Extent Metastatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Max Sung, MD, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 06-0906
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Cancer
Keywords: erlotinib; celecoxib; radiation; progression-free survival
MeSH Terms: conditions — Neoplasms | interventions — Sunitinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Participants treated with chemotherapy and radiotherapy
  Interventions: Drug: sunitinib malate (Sutent); Procedure: radiotherapy

INTERVENTIONS:
Drug: sunitinib malate (Sutent) — Sutent administered PO QD from days 1 to 28 Two weeks after completion of any chemotherapy, maintenance Sutent in 6 week cycles (consisting of Sutent 50 mg PO QD weeks 1-4 followed by no treatment weeks 5-6) until progression or death If no chemotherapy is planned, maintenance Sutent (as described above) will start on day 43.
  Other Names: sunitinib malate; Sutent
Procedure: radiotherapy — Radiation is to be delivered to each site over 10 fractions separated by at least 16 hours. Up to 5 sites may be treated
  Other Names: XRT

SUMMARY:
Cancer is the second leading cause of death in the United States, with approximately 90% of deaths resulting from patients with metastatic spread. Save for notable exceptions such as testicular cancer, chemotherapy alone cannot cure patients with metastases. Some patients with limited metastatic deposits (most commonly colon cancer spread to the liver) can be cured with surgery followed by chemotherapy. Therefore, some patients with metastases should be considered for aggressive local therapy (surgery and/or radiation).

Even though chemotherapy has improved significantly, patients treated with conventional chemotherapy and/or biologically targeted therapy are not cured of their disease. For the most common types of cancer, chemotherapy alone can shrink or stabilize tumors for an average of 6 months before the tumors regrow. Both chemotherapy and biologically targeted therapy have major limitations preventing cure of these patients.

Radiation therapy is an effective modality of treating cancer. Until recently, radiation for metastases was used only to relieve symptoms resulting from local tumor growth. Technological advances, including stereotactic radiotherapy, allow for radiation to be more precisely delivered to the tumor while sparing nearby normal organs. Stereotactic radiotherapy can completely eradicate local tumors with minimal side effects. Stereotactic radiotherapy has never been combined with drug therapy. Sutent is a new F.D.A. approved cancer therapy that targets tumor blood vessels. It is effective against two types of cancer that rarely respond to chemotherapy (GI stromal tumors and kidney cancer). We propose combining biologically targeted drug therapy with physically targeted stereotactic radiotherapy. Our goal is to determine if this is a safe regimen and the best method of combining these treatments. Ultimately, our goal is to cure some patients with previously incurable metastatic cancer with this combination.

ELIGIBILITY:
Inclusion Criteria:

* Zubrod Performance Scale 0-1
* Metastatic disease confirmed by biopsy or imaging
* 5 or fewer sites of metastatic disease on tumor staging (either CT chest/abdomen/pelvis plus bone scan or whole body FDG-PET)
* All tumors measure < 6 cm
* Age > 18
* Chemotherapy must be completed at least 2 weeks prior to radiation
* Signed informed consent
* Adequate bone marrow function, defined as follows;

  1. Platelets > 100,000 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to registration on study
  2. Absolute neutrophil count (ANC) > 1,800 cells/mm3 based on CBC/differential obtained within 2 weeks prior to registration on study
  3. Hemoglobin > 8.0 g/dl based upon CBC/differential obtained within 2 weeks prior to registration on study (Note: The use of transfusion or other intervention to achieve Hgb > 8.0 g/dt is acceptable.)

Exclusion Criteria:

* Other coexisting malignancies or malignancies diagnosed within the previous 3 years with the exception of basal cell carcinoma, cervical carcinoma in situ, and other treated malignancies with no evidence of disease for at least 3 years
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements
* Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF are excluded. The exclusion of patients with active coronary heart disease will be at the discretion of the attending physician.
* Patients with exudative, bloody, or cytologically malignant effusions are not eligible.
* Pregnancy or breast feeding (Women of child-bearing potential are eligible, but must consent to using effective contraception during therapy and for at least 3 months after completing therapy)
* Patients must have no uncontrolled active infection other than that not curable without treatment of their cancer.
* Prior radiation to target area
* Patient may not be receiving any other investigational agents during radiotherapy.
* Prior history of non-inducible bleeding (12/16/09).
* Requirement for continuation of anticoagulation (defined as Coumadin, lovenox, heparin, plavix, aspirin, NSAIDs or similar drugs) during treatment (12/16/09)
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Sung, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Kao J, Packer S, Vu HL, Schwartz ME, Sung MW, Stock RG, Lo YC, Huang D, Chen SH, Cesaretti JA. Phase 1 study of concurrent sunitinib and image-guided radiotherapy followed by maintenance sunitinib for patients with oligometastases: acute toxicity and preliminary response. Cancer. 2009 Aug 1;115(15):3571-80. doi: 10.1002/cncr.24412. PMID 19536893
- [Result] Tong CC, Ko EC, Sung MW, Cesaretti JA, Stock RG, Packer SH, Forsythe K, Genden EM, Schwartz M, Lau KH, Galsky M, Ozao-Choy J, Chen SH, Kao J. Phase II trial of concurrent sunitinib and image-guided radiotherapy for oligometastases. PLoS One. 2012;7(6):e36979. doi: 10.1371/journal.pone.0036979. Epub 2012 Jun 27. PMID 22761653
- [Result] Kao J, Chen CT, Tong CC, Packer SH, Schwartz M, Chen SH, Sung MW. Concurrent sunitinib and stereotactic body radiotherapy for patients with oligometastases: final report of a prospective clinical trial. Target Oncol. 2014 Jun;9(2):145-53. doi: 10.1007/s11523-013-0280-y. Epub 2013 May 10. PMID 23660867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period began January 2007 and was open for recruitment through July 2014 with 47 patients enrolled in the study between February 2007 and September 2010.
Pre-assignment Details: One patient withdrew prior to starting treatment and was excluded from analysis.
  Phase 1: 21 patients in Phase 1 in dose-escalating study to find maximum-tolerated dose Phase 2: 25 patients on the recommended phase II dose, 37.5mg
Groups:
- Advanced Solid Tumor Malignancy: Patients were eligible if they had histologically or cytological documented advanced solid tumor malignancy with radiographic evidence of 1 to 5 sites of active metastatic disease.
Period: Phase 1-Radiation 40 Gy + Sunitinib 25mg
Arm/Group | Advanced Solid Tumor Malignancy
Started | 3
Completed | 3
Not Completed | 0
Period: Phase 1-Radiation 40 Gy+Sunitinib 37.5mg
Arm/Group | Advanced Solid Tumor Malignancy
Started | 3
Completed | 3
Not Completed | 0
Period: Phase 1-Radiation 50 Gy+Sunitinib 37.5mg
Arm/Group | Advanced Solid Tumor Malignancy
Started | 10
Completed | 10
Not Completed | 0
Period: Phase 1-Radiation 50Gy +Sunitinib 50mg
Arm/Group | Advanced Solid Tumor Malignancy
Started | 5
Completed | 0
Not Completed | 5
Not completed — acute toxicity | 5
Period: Phase 2-Radiation 50Gy +Sunitinib 37.5mg
Arm/Group | Advanced Solid Tumor Malignancy
Started | 26 (Not all patients participated in both Phase 1 and Phase II)
Completed | 25
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: N=21 participants Patients enrolled between Feb 2007 and May 2008
- Phase II Advanced Solid Tumor Malignancy: Patients were eligible if they had histologically or cytological documented advanced solid tumor malignancy with radiographic evidence of 1 to 5 sites of active metastatic disease.
  N=26 participants Patients enrolled between February 2008 and September 2010
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II Advanced Solid Tumor Malignancy | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Continuous [Median (Full Range); unit: years] | 65 [47 to 82] | 63 [54 to 83] | 64 [47 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 14 | 18 | 32
ECOG Performance status [Number; unit: participants] — ECOG performance status is an attempt to quantify cancer patients' general well-being and activities of daily life.
  0 Fully active, able to carry on all predisease activities with restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Out of bed > 50%
  3. Capable of only limited self-care , confined to bed or chair > 50% waking hours
  4. Completely disabled, cannot carry on any self-care, totally confined to bed or chair
  participants
    0 | 7 | 4 | 11
    1 | 9 | 13 | 22
    2 | 5 | 8 | 13
Prior systemic chemotherapy [Number; unit: participants]
  Yes | 13 | 11 | 24
  No | 8 | 14 | 22
Prior radiation therapy [Number; unit: participants]
  Yes | 11 | 10 | 21
  No | 10 | 15 | 25
Number of metastases [Number; unit: participants]
  1 | 13 | 13 | 26
  2 | 3 | 5 | 8
  >=3 | 5 | 7 | 12
Largest Tumor size [Number; unit: participants]
  <=3cm | 11 | 15 | 26
  >=3cm | 10 | 10 | 20
Number of involved organs [Number; unit: participants]
  1 | 17 | 14 | 31
  >=2 | 4 | 11 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: Sunitinib (SU) and radiation (IGRT) doses were sequentially escalated using a ping-pong strategy according to a 3 + 3 design phase 1 study. The starting dose was sunitinib 25 mg and IGRT 40 Gy. MTD reflects the highest dose that did not cause a dose limiting toxicity. Toxicity was in assessed in patients at regular intervals by using the Common Terminology Criteria for Adverse Events criteria (version 3.0). Dose limiting events were defined as any grade 4 or 5 toxicity and unexpected grade 3 toxicity. Expected grade 3 toxicities from radiation include mucositis or esophagitis lasting ≤7 days. Grade 3 metabolic and hematologic toxicities are considered expected events with sunitinib and therefore were not considered DLTs
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Radiation 40Gy + Sunitinib 25 mg | Phase 1 - Radiation 40Gy + Suniitnib 37.5 mg | Phase 1 - Radiation 50Gy + Sunitinib 37.5mg | Phase 1 - Radiation 50Gy + Sunitinib 50mg
Number analyzed (Participants) | 3 | 3 | 10 | 5
Participants | 0 | 0 | 1 | 2

2. Primary Outcome: Number of Participants With Particular Disease Status
Description: Number of participants who have no evidence of disease and number of participants with distant metastases.
Time Frame: 5 years
Population: Phase 2 only
Measure: Number; unit: participants
Arm/Group | Advanced Solid Tumor Malignancy
Number analyzed (Participants) | 46
participants
  No evidence of disease | 12
  distant metastases | 3

3. Secondary Outcome: Percentage of Patients With Toxicity Grade 3 or Higher
Description: % of patients experienced one or more grade ≥ 3 toxicities. Toxicity is graded as mild (Grade 1), moderate (Grade 2), severe (Grade 3), or life-threatening (Grade 4),and death (Grade 5).
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Solid Tumor Malignancy
Number analyzed (Participants) | 46
Participants | 15

4. Secondary Outcome: Percentage of Patients With Local Control
Description: Local control was defined as a tumor volume equal to or less than the tumor volume at start of radiotherapy.
Time Frame: 4 years
Population: the 4-year estimates for local control
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Advanced Solid Tumor Malignancy
Number analyzed (Participants) | 46
percentage of participants | 75 [55 to 87]

5. Secondary Outcome: Percentage of Patients With Distant Control
Description: Distant control defined as distant metastasis contained outside of the radiation field within months of treatment.
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Advanced Solid Tumor Malignancy
Number analyzed (Participants) | 46
percentage of participants | 40 [24 to 55]

6. Secondary Outcome: Quality of Life
Time Frame: 4-6 weeks after radiation therapy
Population: data not collected
Arm/Group | Advanced Solid Tumor Malignancy
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants According Failure and Survival
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Solid Tumor Malignancy
Number analyzed (Participants) | 46
Participants
  alive without evidence of disease | 12
  alive with distant metastases | 3
  dead from distant metasteses | 22
  dead from local progression | 1
  dead from comorbid illness | 6
  dead from treatment-related toxicities | 2

ADVERSE EVENTS:
Time Frame: Patients from Phase I and patients from Phase II, various doses of sunitinib (25mg to 50mg) and radiotherapy (40 to 50Gy). Median follow up was 3.6 years. Patients were followed until death.
Groups:
- Phase 1: N=21 participants Patients enrolled between Feb 2007 and May 2008
- Phase 2: Patients were eligible if they had histologically or cytological documented advanced solid tumor malignancy with radiographic evidence of 1 to 5 sites of active metastatic disease.
  N=26 participants Patients enrolled between February 2008 and September 2010
Arm/Group | Phase 1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 13/21 | 18/26
Serious Adverse Events (participants affected / at risk) | 13/21 | 13/26
Other Adverse Events (participants affected / at risk) | 21/21 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=21) | Phase 2 (N=26)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Immune system disorders) | 4 | 2
LFT abnormalities (Hepatobiliary disorders) | 3 | 1 — liver function test
Thrombocytopenia (Immune system disorders) | 3 | 4
Bleeding (Blood and lymphatic system disorders) | 1 | 2
Metabolic abnormalities (Endocrine disorders) | 2 | 1
Increased creatinine (Renal and urinary disorders) | 0 | 1
Nausea/vomiting (General disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 13 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=21) | Phase 2 (N=26)
Anemia (Blood and lymphatic system disorders) | 14 | 16
Neutropenia (Blood and lymphatic system disorders) | 12 | 12
Fatigue (General disorders) | 13 | 18
LFT abnormalities (Hepatobiliary disorders) | 8 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 11
Mucositis/stomatitis (Infections and infestations) | 7 | 8
Nausea/vomiting (General disorders) | 6 | 7
Skin changes (Skin and subcutaneous tissue disorders) | 4 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 5
Hypertension (Cardiac disorders) | 3 | 3
Bleeding (Blood and lymphatic system disorders) | 0 | 2
Metabolic abnormalities (Metabolism and nutrition disorders) | 3 | 1
Increased creatinine (Renal and urinary disorders) | 0 | 5
Hand foot syndrome (Infections and infestations) | 2 | 0
Hypothryrodism (Metabolism and nutrition disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes